CLINICAL TRIAL: NCT02678325
Title: Tolerance of Early High Protein Nutrition of the Critically Ill: Comparison of a Protein-rich Enteral Formula With a Standardized High Carbohydrate Product on Total Calorie and Protein Intake
Brief Title: The Basel Enteral High Protein Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2016-00041
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: High Enteral Protein Nutrition; Muscle Breakdown; Autophagy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized normal protein enteral nutrition formula (Active Comparator): Standardized enteral nutrition formula with a caloric density of 1.2 kcal/ml and protein percentage 20% of the total caloric intake
  Interventions: Other: Standardized normal protein enteral nutrition
- Standardized high protein enteral nutrition formula (Experimental): Standardized enteral nutrition formula with a caloric density of 1.2 kcal/ml and protein percentage 33% of the total caloric intake
  Interventions: Other: Standardized high protein enteral nutrition

INTERVENTIONS:
Other: Standardized high protein enteral nutrition — A double-blind randomized controlled clinical trial of critically ill patients to explore values of high enteral protein administration on muscle breakdown and mortality.
  Arms: Standardized high protein enteral nutrition formula
Other: Standardized normal protein enteral nutrition — double-blind randomized controlled clinical trial of critically ill patients to explore values of high enteral protein administration (compared to normal enteral protein administration) on muscle breakdown and mortality.
  Arms: Standardized normal protein enteral nutrition formula

SUMMARY:
The objective of this study is to compare the difference in daily protein intake of critically ill patients in two standardized enteral nutrition formulas (20% versus 33% percent) with the same caloric density of 1.2 kcal/ml.

The total amount of protein taken in on day four after starting the early enteral feeding is defined as primary endpoint.

DETAILED DESCRIPTION:
For years, the Surgical Intensive Care Unit of the University Hospital Basel has used an early enteral approach for the feeding of critically ill patients with different formulas that have high protein content (20% of total energy). However, the energy goal in the first week is only 20 kcal for normal-weight and 12.5 kcal for obese patients, which results in daily protein amounts of 0.8 to 1 g/kg bodyweight (BW), so that additional protein has to be administered. Due to a suggestion of the dietetic service of the University Hospital Basel, Fresenius Kabi produced a whey based enteral feeding formula for intensive care patients. Specific further adaptations for this patient group included micronutrients and a fatty acid profile as well as low fibres. Surgical Intensive Care Unit of the University Hospital Basel now are offered the opportunity to test this formula in clinical practice and hypothesize that this specific high-protein (30% of energy) enteral formula reaches the same amount of daily caloric intake with a higher total daily amount of protein and equal intestinal tolerance compared to a usual intestinal nutritional formula.

In order to test this hypothesis, investigators plan a double-blind, randomized and controlled study with the aim to achieve a target protein quantity of ≥1.3 g/kg BW with an energy target of 20kcal/kg BW per day, based on a new, specifically designed formula for critically ill patients. The amount of protein on day four after starting the early enteral feeding is defined as primary endpoint. Secondary endpoints are the total amount of calories, the nitrogen balance on day five as well as side effects like gastric residual content, diarrhoea and constipation. Inclusion criteria were an expected stay at the ICU of four days or longer on admission and 18 years of age or older Exclusion criteria consisted of BMI ≤ 18, pregnancy, intestinal perforation, mechanical intestinal obstruction, terminal state of consuming disease, severely impaired liver function and noradrenaline ≥0.5µg/kg BW/min.. On this purpose, 90 critically ill patients will get either of the two enteral feeding products as described above. In case of the event that an increased protein intake can be obtained by the protein-rich formula, an additional study will investigate the influence of early protein-rich nutrition on skeletal muscle wasting with critically ill patients.

In a pre-study investigators will administer the high protein formula to 20 patients to test tolerance and suitability for the nutritional Targets in question. Tolerance will be defined by the absence of one of the following clinical symptoms :

* Reflux
* Diarrhoea
* Constipation
* Nausea
* Vomiting

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 years or older)
* expected stay at the ICU of four days upon admittance or longer
* expected enteral feeding during at least four days.

Exclusion Criteria:

* BMI ≤ 18
* Mechanical intestinal obstruction
* Intestinal perforation
* Severely impaired liver function
* Terminal state of consuming disease
* Noradrenaline ≥0.5µg/kg BW/min
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-05-21 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The amount of protein | 4 days
  The amount of protein administered on day four after starting the early enteral feeding.

SECONDARY OUTCOMES:
The total amount of calories | 4 days
  Indirect Calorimetry
The nitrogen balance on day four | 4 days
  Nitrogen input - nitrogen loss measured over 4 days
Gastric residual Content in ml | 4 days
  ml
Number of diarrhea events | 4 days
  Number
occurence of constipation as measured in time without defecation | 4 days
  time frame without defecation

CONTACTS AND LOCATIONS:
Overall Officials: Martin Siegemund, Prof. Dr. MD, Study Director — Deputy Chief Physician, Surgical Intensive Care Unit, University Hospital Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tedeschi-Jockers F, Reinhold S, Hollinger A, Tuchscherer D, Kiss C, Gantner L, Ledergerber K, Zimmermann S, Scheuzger J, Huber J, Siegemund M. A new high protein-to-energy enteral formula with a whey protein hydrolysate to achieve protein targets in critically ill patients: a prospective observational tolerability study. Eur J Clin Nutr. 2022 Mar;76(3):419-427. doi: 10.1038/s41430-021-00956-9. Epub 2021 Jun 24. PMID 34168292